CLINICAL TRIAL: NCT03916965
Title: Prospective Observational Cohort Study in Patients With SIDSMA Treated With Stents
Brief Title: Stent Implantation for Patients With SIDSMA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.62
Record Dates: First submitted 2019-04-07; First posted 2019-04-16 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-02

CONDITIONS: Dissection of the Superior Mesenteric Artery
Keywords: dissection of the superior mesenteric artery; patency of stents; remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the prognosis in patients with spontaneous isolated dissection of the superior mesenteric artery (SIDSMA) who have been treated with stents.

DETAILED DESCRIPTION:
This study is a prospective, observational study. Patients who have been diagnosed as spontaneous isolated dissection of the superior mesenteric artery (SIDSMA) and treated with stents are enrolled in the study. We will evaluate the patency of stent, remodeling of the dissection and the relief of the symptoms in the next 1 years after patients have received stents.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female over 18 years of age
2. Diagnosed as spontaneous isolated dissection of the superior mesenteric artery
3. Patients have been successfully treated with stents
4. Patients are willing to participate in this study

Exclusion Criteria:

1. Life expectancy of < 5 years;
2. Other surgeries or endovascular treatments have been taken concurrently.
3. Elevated serum level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed as spontaneous isolated dissection of the superior mesenteric artery (SIDSMA) and treated with stents are potential candidates for the study. All participants must meet all inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Patency of stents deployed in the superior mesenteric artery | 12 months post-procedure
  The patency of stents deployed in the superior mesenteric artery shall be evaluated via computed tomographic angiography
Remodeling of the superior mesenteric artery | 12 months post-procedure
  Complete remodeling was defined as the absence of residual arterial dissection and stenosis via follow-up computed tomographic angiography. Incomplete remodeling was defined as improved luminal patency of the superior mesenteric artery but worse than complete remodeling.

SECONDARY OUTCOMES:
Relief of symptoms | 12 months post-procedure
  Most of patients with SIDSMA are symptomatic. The symptoms mainly include abdominal pain, hematochezia, nausea and vomiting.After the procedure, the time delay between the stent implantation and disappearance of these symptoms are documented.
Recurrence | 12 months post-procedure
  New dissection in the superior mesenteric artery

CONTACTS AND LOCATIONS:
Overall Officials: Ziheng Wu, Principal Investigator — Zhejiang University
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Qiu C, Wu Z, He Y, Tian L, Zhu Q, Shang T, Zhang H, Li D. Endovascular therapy versus medical treatment for spontaneous isolated dissection of the superior mesenteric artery. Cochrane Database Syst Rev. 2022 Sep 8;9(9):CD014703. doi: 10.1002/14651858.CD014703.pub2. PMID 36074662